CLINICAL TRIAL: NCT04588259
Title: Efficacy and Safety of Fast-acting Insulin Aspart Compared to NovoRapid® Both in Combination With Insulin Degludec With or Without Metformin in Adults With Diabetes
Brief Title: Research Study to Compare a New Medicine "Fast-acting Insulin Aspart" to Another Medicine "Insulin Aspart" in Chinese People With Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1218-4357; U1111-1197-8289 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faster aspart (Experimental): 4 daily injections of faster aspart given with insulin degludec and with or without metformin
  Interventions: Drug: Faster aspart; Drug: Insulin degludec
- Insulin aspart (Active Comparator): 4 daily injections of insulin aspart given with insulin degludec and with or without metformin
  Interventions: Drug: Insulin aspart; Drug: Insulin degludec

INTERVENTIONS:
Drug: Faster aspart — Administered s.c. (subcutaneously, under the skin) for 16 weeks
  Arms: Faster aspart
Drug: Insulin aspart — Administered s.c. (subcutaneously, under the skin) for 16 weeks
  Arms: Insulin aspart
Drug: Insulin degludec — Administered s.c. (subcutaneously, under the skin) for 16 weeks

SUMMARY:
Fast-acting insulin aspart (faster aspart) will be tested to see how well it works and if it is safe. The study compares 2 medicines for type 1 and type 2 diabetes - faster aspart (a new medicine) and insulin aspart (a medicine doctors can already prescribe). Participants will either get faster aspart or insulin aspart (NovoRapid®) - which treatment is decided by chance. Both medicines will be taken together with insulin degludec. Participants will need to take 1 injection 4 times every day: 3 injections 0-2 minutes before breakfast, lunch and dinner and 1 injection at the same time every day. All study medicines are provided in pens. A pen is a tool to inject insulin under the skin.The study will last for about 7 months (30 weeks). Participants will have 11 clinic visits and 17 phone contacts with the study doctor. At 8 clinic visits participants will have blood samples taken. At 3 clinic visits participants cannot eat or drink (water is allowed) 8 hours before the visits - at 2 of these visits participants will be asked to drink a liquid meal and to stay at the clinic for about 5 hours. Participants will fill in a diary the last 3 days before the visits/phone contacts. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age above or equal to 18 years at the time of signing informed consent
* Diagnosed with Diabetes Mellitus, Type 1 (T1DM) at least or equal to 1 year prior to screening or diagnosed with Diabetes Mellitus, Type 2 (T2DM) at least or equal to 5 years prior to screening
* Treated with a basal-bolus insulin regimen or a premix insulin regimen at least or equal to 1 year prior to screening. Insulin regimen must be unchanged within 60 days prior to screening. A basal-bolus insulin regimen is defined as basal insulin once or twice daily and bolus insulin taken with meals at least thrice daily. A premix insulin regimen is defined as premix insulin twice or thrice daily
* For subjects with T1DM: not treated with any oral anti-diabetes drugs (OADs) for at least 90 days prior to screening. For subjects with T2DM: not treated with any OADs or treated with 1-2 OADs within 90 days prior to screening. Allowed OADs are metformin, alpha-glucosidase inhibitor, sodium-glucose co-transporter-2 inhibitors (SGLT2i) and dipeptidyl peptidase-4 inhibitors (DPP4i). Change in OAD and dose prior to screening is allowed.
* HbA1c 7.5-9.5% (both inclusive) as assessed by central laboratory at screening

Exclusion Criteria:

* Any of the following: myocardial infarction, stroke, hospitalisation for unstable angina pectoris or transient ischaemic attack within the past 180 days prior to the day of screening
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within the past 90 days prior to the day of screening
* Anticipated initiation or change in concomitant medications (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or corticosteroids)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (Dept. 1452), Study Director — Novo Nordisk A/S
Locations (40):
- China (38):
  - Anhui Provincial Hospital-Endocrinology, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University-Endocrinology, Hefei, Anhui
  - Beijing Chao-Yang Hospital, Capital Medical University-Endocrinology, Beijing, Beijing Municipality
  - The Fifth Medical Center of PLA General Hospital-Endocrinology, Beijing, Beijing Municipality
  - The General Hospital of the PLA Rocket Force-Endocrinology, Beijing, Beijing Municipality
  - Chinese People's Liberation Army General Hospital-Endocrinology, Beijing, Beijing Municipality
  - Beijing Pinggu Hospital-Endocrinology, Beijing, Beijing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Shantou University Medical College-Endocrinology, Shantou, Guangdong
  - The Second Affiliated Hospital of Guangxi Medical University-Endocrinology, Nanning, Guangxi
  - Cangzhou People's Hospital-Endocrinology, Cangzhou, Hebei
  - Hengshui People's Hospital (Harrison International Peace Hospital)-Endocrinology, Hengshui, Hebei
  - The Second Hospital of Hebei Medical University-Endocrinology, Shijiazhuang, Hebei
  - Tangshan Gongren Hospital-Endocrinology, Tangshan, Hebei
  - Yueyang Central Hospital-Endocrinology, Yueyang, Hunan
  - Inner Mongolia People's Hospital-Endocrinology, Hohhot, Inner Mongolia
  - The affiliated Hospital of Inner Mongolia Medical University-Endocrinology, Hohhot, Inner Mongolia
  - Changzhou No.2 People's Hospital, Yanghu Branch, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University-Endocrinology, Nanjing, Jiangsu
  - Jiangsu Province Hospital-Endocrinology, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital-Endocrinology, Nanjing, Jiangsu
  - Suzhou Municipal Hospital-Endocrinology, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Jiangsu University-Endocrinology, Zhenjiang, Jiangsu
  - Jiangxi Provincial People's Hospital-Endocrinology, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University-Endocrinology, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Bethune hospital of Jilin University-Endocrinology, Changchun, Jilin
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong
  - Shanghai Tenth People's Hospital (Tenth People's of Tongji University)-Endocrinology, Shanghai, Shanghai Municipality
  - Shanghai Fifth People's Hospital-Endocrinology, Shanghai, Shanghai Municipality
  - Central Hospital of Minhang District, Shanghai-Endocrinology, Shanghai, Shanghai Municipality
  - General Hospital of Tianjin Medical University-Endocrinology, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University-Endocrinology, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province-Endocrinology, Kunming, Yunnan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
- Hong Kong (2):
  - Master Centre for Hong Kong, Kowloon
  - Prince of Wales Hospital, Shatin, New Territories

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 31 sites in China.
Pre-assignment Details: The trial included an 8-week run-in period and a 16-week treatment period. During the run-in period, participants received NovoRapid both in combination with insulin degludec with or without metformin primarily for optimisation of the basal insulin treatment. Participants were then randomised 1:1 to receive either 'Faster aspart + insulin degludec with or without metformin' or 'NovoRapid + insulin degludec with or without metformin' during the treatment period.
Groups:
- Faster aspart: Participants received subcutaneous injections of NovoRapid + insulin degludec with or without metformin for 8 weeks in the run-in period, followed by Faster aspart + insulin degludec with or without metformin subcutaneously for 16 weeks in the treatment period. During the run-in period, insulin degludec dose was adjusted weekly by the investigator based on the mean of three pre-breakfast self-measured plasma glucose (SMPG) values measured on the last two days prior to and on the day of contact. If one of the SMPG values were below target (less than 4.0 millimole per litre (mmol/L) or 71 milligrams per decilitre (mg/dL)) then the insulin degludec dose was adjusted according to the titration guideline specified in the protocol. Faster aspart was titrated from randomisation (week 0) and onwards, twice weekly to reach the glycaemic target of pre-prandial and bedtime plasma glucose (PG) between 4.0-6.0 mmol/L (71 - 108 mg/dL) in a treat-to-target fashion.
- NovoRapid: Participants received subcutaneous injections of NovoRapid thrice daily + insulin degludec once daily with or without metformin for 24 weeks (8 weeks run-in period + 16 weeks treatment period). During the run-in period, insulin degludec dose was adjusted weekly by the investigator based on the mean of three pre-breakfast SMPG values measured on the last two days prior to and on the day of contact. If one of the SMPG values were below target (less than 4.0 mmol/L or 71 mg/dL) then the insulin degludec dose was adjusted according to the titration guideline specified in the protocol. NovoRapid was titrated from randomisation (week 0) and onwards, twice weekly to reach the glycaemic target of pre-prandial and bedtime PG between 4.0-6.0 mmol/L (71 - 108 mg/dL) in a treat-to-target fashion.
Period: Run-in period
Arm/Group | Faster aspart | NovoRapid
Started | 0 | 331
Completed | 0 | 300
Not Completed | 0 | 31
Not completed — Run-in failure | 0 | 23
Not completed — Withdrawn before randomisation | 0 | 8
Period: Treatment period
Arm/Group | Faster aspart | NovoRapid
Started | 150 | 150
Full analysis set | 150 | 150
Safety analysis set | 150 | 150
Completed | 144 | 144
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 6 | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) which included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Faster Aspart | NovoRapid | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.79 (10.65) | 55.24 (12.02) | 56.02 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 68 | 136
  Male | 82 | 82 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 149 | 150 | 299
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 150 | 150 | 300
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c) (Percentage [%])
Description: Change from baseline (week 0) in HbA1c (%) as evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Baseline (week 0), week 16
Population: Full analysis set (FAS) which included all randomised participants. Number of participants analysed = Number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 143 | 145
Percentage of HbA1c | -0.57 (0.63) | -0.54 (0.73)
Statistical Analysis 1: Comparison: Faster aspart vs NovoRapid; The outcome measure was analysed using mixed-effect model for repeated measurement (MMRM) where all calculated changes in HbA1c from baseline at visits were included in analysis. Model included treatment and stratification of type 1 diabetes mellitus/ type 2 diabetes mellitus (T1DM/T2DM) as fixed factors, HbA1c at baseline as covariate and interactions between all fixed factors and visit. An unstructured covariance matrix described the variability for the repeated measurements for a participant; Test type: Non-Inferiority — The upper limit of the 95% confidence interval (CI) for the difference between faster aspart and NovoRapid was compared to a non-inferiority margin of 0.4%. If it was below or equal to 0.4%, non-inferiority was considered to be established and effect demonstrated; p = 0.5102, Mixed Models Analysis — p-values are from the 2-sided test for treatment difference evaluated at the 5% level; Treatment difference = -0.05, 95% CI 2-sided [-0.19 to 0.09]

2. Primary Outcome: Change From Baseline in HbA1c (Millimoles Per Mole [mmol/Mol])
Description: Change from baseline (week 0) in HbA1c (mmol/mol) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Baseline (week 0), week 16
Population: FAS which included all randomised participants. Number of participants analysed = Number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 143 | 145
mmol/mol | -6.18 (6.84) | -5.89 (7.94)
Statistical Analysis 1: Comparison: Faster aspart vs NovoRapid; The outcome measure was analysed using a mixed-effect model for repeated measurements (MMRM) where all calculated changes in HbA1c from baseline at visits are included in the analysis. The model includes treatment and stratification (T1DM/T2DM) as fixed factors, HbA1c at baseline as covariate and interactions between all fixed factors and visit. An unstructured covariance matrix is used to describe the variability for the repeated measurements for a participant; Test type: Non-Inferiority — The upper limit of the 95% CI for the difference between faster aspart and NovoRapid was compared to a non-inferiority margin of 0.4%. If it was below or equal to 0.4%, non-inferiority was considered to be established and effect demonstrated; p = 0.5102, Mixed Models Analysis — p-values are from the 2-sided test for treatment difference evaluated at the 5% level; Treatment Difference = -0.52, 95% CI 2-sided [-2.08 to 1.03]

3. Secondary Outcome: Change From Baseline in 30-minutes, 1-hour, 2-hour and 3-hour Post Prandial Glucose (PPG) Increment (Meal Test)
Description: Change from baseline (week 0) in 30-minute, 1-hour, 2-hour and 3-hour PPG increment (meal test) was evaluated at 16 weeks. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. Meal test: The participants were given a carbohydrate-rich standardised liquid meal immediately after bolus (faster aspart or NovoRapid) infusion in the morning of the meal test. The participants were to consume the meal as quickly as possible (within 12 minutes) and blood samples were drawn after 30 minutes, 1, 2 and 3 hours from the start of the meal. PPG incremental value for each time point was derived as PPG value at that time point minus the preprandial glucose value.
Time Frame: Baseline (week 0), week 16 (30 minutes, 1 hour, 2 hour and 3 hour)
Population: FAS which included all randomised participants. Number of participants analysed = Number of participants contributed to the analysis and Number analysed = Number of participants evaluable for each timepoint.
Measure: Mean (Standard Deviation); unit: Millimoles per litre (mmol/L)
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 144 | 146
Millimoles per litre (mmol/L)
  30-min: number analyzed (Participants) | 143 | 146
  30-min | -1.01 (2.31) | 0.18 (2.15)
  1-hour | -0.94 (3.08) | 0.46 (3.00)
  2-hour: number analyzed (Participants) | 144 | 145
  2-hour | 0.21 (4.16) | 0.64 (4.05)
  3-hour: number analyzed (Participants) | 144 | 144
  3-hour | 0.77 (4.01) | 0.65 (4.55)

4. Secondary Outcome: Change From Baseline in 30-minutes, 1-hour, 2-hour and 3-hour PPG (Meal Test)
Description: Change from baseline (week 0) in 30-minute, 1-hour, 2-hour and 3-hour PPG (meal test) was evaluated at 16 weeks. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. Meal test: The participants were given a carbohydrate-rich standardised liquid meal immediately after bolus (faster aspart or NovoRapid) infusion in the morning of the meal test. The participants were to consume the meal as quickly as possible (within 12 minutes) and blood samples were drawn after 30 minutes, 1, 2 and 3 hours from the start of the meal.
Time Frame: Baseline (week 0), week 16 (30 minutes, 1 hour, 2 hour and 3 hour)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 144 | 146
mmol/L
  30-min: number analyzed (Participants) | 143 | 146
  30-min | -0.64 (3.06) | 0.37 (2.67)
  1-hour | -0.55 (3.53) | 0.64 (3.10)
  2-hour: number analyzed (Participants) | 144 | 145
  2-hour | 0.60 (4.53) | 0.81 (4.16)
  3-hour: number analyzed (Participants) | 144 | 144
  3-hour | 1.16 (4.41) | 0.87 (4.55)

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in fasting plasma glucose (FPG) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Baseline (week 0), week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 143 | 145
mmol/L | 0.39 (2.50) | 0.20 (2.11)

6. Secondary Outcome: Change From Baseline in 7-9-7-point Self-measured Plasma Glucose (SMPG) for Mean of the 7-9-7-point Profile
Description: Change from baseline (week 0) in mean of the 7-9-7 point SMPG profile was evaluated after 16 weeks of randomisation. 7-9-7 SMPG point profile was performed on the 3 consecutive days just before selected visit. 7-point profile (day 3 and day 1 before selected visit): before breakfast, 60 minutes after the start of breakfast, before lunch, 60 minutes after the start of lunch, before main evening meal, 60 minutes after the start of main evening meal, and at bedtime. 9-point profile (day 2 before selected visit) included all timepoints of 7-points profile with addition of SMPG measurement at 4 a.m. and before breakfast on the following day. The mean of the 7-9-7-point profile was defined as the area under the curve profile divided by the measurement time, and was calculated using the linear trapezoidal technique. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Baseline (week 0), week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 144 | 144
mmol/L | -0.73 (1.55) | -0.76 (1.78)

7. Secondary Outcome: Change From Baseline in 7-9-7-point SMPG for 1-hour PPG (Mean, Breakfast, Lunch, Main Evening Meal)
Description: Change from baseline (week 0) in 1-hour PPG (breakfast, lunch, main evening meal and mean over all meals) of the 7-9-7 point SMPG profile was evaluated after 16 weeks of randomisation. 7-9-7 SMPG point profile was performed on the 3 consecutive days just before selected visit. 7-point profile (day 3 and day 1 before selected visit): before breakfast, 60 minutes after the start of breakfast, before lunch, 60 minutes after the start of lunch, before main evening meal, 60 minutes after the start of main evening meal, and at bedtime. 9-point profile (day 2 before selected visit) included all timepoints of 7-points profile with addition of SMPG measurement at 4 a.m. and before breakfast on the following day. Results were derived from the three profiles: post-breakfast, post-lunch, post-main evening meal. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Baseline (week 0), week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 142 | 140
mmol/L
  1 hour after breakfast: number analyzed (Participants) | 139 | 139
  1 hour after breakfast | -1.01 (2.38) | -0.37 (2.85)
  1 hour after lunch: number analyzed (Participants) | 141 | 138
  1 hour after lunch | -1.16 (2.62) | -1.07 (2.65)
  1 hour after main evening meal: number analyzed (Participants) | 142 | 138
  1 hour after main evening meal | -1.34 (3.10) | -0.68 (2.68)
  1 hour after all meals | -1.17 (1.92) | -0.70 (2.11)

8. Secondary Outcome: Change From Baseline in 7-9-7-point SMPG for PPG Increment (Mean, Breakfast, Lunch, Main Evening Meal)
Description: Change from baseline (week 0) in PPG increment of the 7-9-7 point SMPG profile was evaluated after 16 weeks of randomisation. 7-9-7 SMPG point profile was performed on the 3 consecutive days just before selected visit. 7-point profile (day 3 and day 1 before selected visit): before breakfast, 60 minutes after the start of breakfast, before lunch, 60 minutes after the start of lunch, before main evening meal, 60 minutes after the start of main evening meal, and at bedtime. 9-point profile (day 2 before selected visit) included all timepoints of 7-points profile with addition of SMPG measurement at 4 a.m. and before breakfast on the following day. PPG increment for each meal was derived from the 7-point and 9-point profile as the difference between PPG values and the PG value before the meal in each separate profile. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Baseline (week 0), week 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 141 | 140
mmol/L
  Breakfast: number analyzed (Participants) | 138 | 139
  Breakfast | -1.37 (2.37) | -0.49 (2.50)
  Lunch: number analyzed (Participants) | 140 | 138
  Lunch | -1.09 (2.89) | -0.19 (2.60)
  Main evening meal: number analyzed (Participants) | 140 | 138
  Main evening meal | -0.34 (2.69) | 0.15 (2.69)
  All meals | -0.95 (1.60) | -0.22 (1.58)

9. Secondary Outcome: Change From Baseline in 7-9-7-point SMPG for Fluctuation in 7-9-7-point Profile: Ratio to Baseline
Description: Fluctuation in SMPG profile was the average absolute difference from the mean of the SMPG profile. Change from baseline is represented as ratio to baseline value. 7-9-7 SMPG point profile was performed on the 3 consecutive days just before selected visit. 7-point profile (day 3 and day 1 before selected visit): before breakfast, 60 minutes after the start of breakfast, before lunch, 60 minutes after the start of lunch, before main evening meal, 60 minutes after the start of main evening meal, and at bedtime. 9-point profile (day 2 before selected visit) included all timepoints of 7-points profile with addition of SMPG measurement at 4 a.m. and before breakfast on the following day. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: Baseline (week 0), week 16
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of 7-9-7-point SMPG
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 144 | 144
Ratio of 7-9-7-point SMPG | 0.77 (55.19) | 0.73 (47.37)

10. Secondary Outcome: Number of Participants Who Achieved HbA1c Less Than (<) 7.0 (Percent [%]) (Yes/No)
Description: Number of participants who achieved HbA1c < 7% measured as 53 mmol/mol at week 16 is presented. In the reported data, "Yes" infers the number of participants who have achieved HbA1c values < 7% and "No" infers the number of participants who have not achieved HbA1c values < 7%. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: At week 16
Population: FAS which included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Participants
  Yes | 59 | 55
  No | 91 | 95

11. Secondary Outcome: Number of Participants Who Achieved HbA1c <7.0% Without Severe Hypoglycaemia Episodes (Yes/No)
Description: Number of participants who achieved HbA1c < 7% (measured as 53 mmol/mol) without severe hypoglycaemia episodes at week 16 is presented. In the reported data, "Yes" infers the number of participants who have achieved HbA1c values < 7% without severe hypoglycaemia episodes and "No" infers the number of participants who have not achieved HbA1c values less than the 7%. without severe hypoglycaemia episodes The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: At week 16
Population: FAS which included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Participants
  Yes | 59 | 55
  No | 91 | 95

12. Secondary Outcome: Number of Participants Who Achieved PPG Target (Overall Mean of Daily PPG Measurements in SMPG) for Overall PPG (1-hour) Less Than or Equal (≤) to 7.8 mmol/L (Yes/No)
Description: Number of participants who achieved overall PPG (1-hour) ≤ 7.8 mmol/L measured as 140 milligrams per deciliter (mg/dL) at week 16 is presented. In the reported data, "Yes" infers the number of participants who have achieved overall PPG (1-hour) values ≤ 7.8 mmol/L and "No" infers the number of participants who have not achieved overall PPG (1-hour) values ≤ 7.8 mmol/L. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: At week 16
Population: FAS which included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Participants
  Yes | 61 | 51
  No | 89 | 99

13. Secondary Outcome: Number of Participants Who Achieved PPG Target (Overall Mean of Daily PPG Measurements in SMPG) for Overall PPG (1-hour) Less Than or Equal (≤) to 7.8 mmol/L Without Severe Hypoglycaemia (Yes/No)
Description: Number of participants who achieved overall PPG (1-hour) ≤ 7.8 mmol/L (measured as 140 mg/dL) without severe hypoglycaemia at week 16 is presented. In the reported data, "Yes" infers the number of participants who have achieved overall PPG (1-hour) values ≤ 7.8 mmol/L without severe hypoglycaemia and "No" infers the number of participants who have not achieved overall PPG (1-hour) values ≤ 7.8 mmol/L without severe hypoglycaemia. The results are based on the last in-trial value, which included the last available measurement in the in-trial period.
Time Frame: At week 16
Population: FAS which included all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Participants
  Yes | 61 | 51
  No | 89 | 99

14. Secondary Outcome: Insulin Dose (Units/Day): Total Basal
Description: Total basal insulin dose was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: At week 16
Population: Safety analysis set (SAS) which included all participants receiving at least one dose of randomised treatment. Number of participants analysed = Number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Units/day
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 144 | 144
Units/day | 27.01 (14.37) | 27.21 (13.30)

15. Secondary Outcome: Insulin Dose (Units/Day): Total Bolus
Description: Total bolus insulin dose was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: At week 16
Population: SAS which included all participants receiving at least one dose of randomised treatment. Number of participants analysed = Number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Units/day
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 144 | 144
Units/day | 39.49 (17.08) | 39.16 (16.90)

16. Secondary Outcome: Insulin Dose (Units/Day): Individual Meal Insulin Dose
Description: Individual meal time bolus insulin dose for breakast, lunch and main evening meal was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: At week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units/day
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 144 | 144
Units/day
  Breakfast | 12.00 (5.90) | 11.54 (6.12)
  Lunch | 13.67 (6.02) | 13.84 (6.11)
  Main evening meal | 13.82 (6.38) | 13.78 (5.89)

17. Secondary Outcome: Insulin Dose (Units/kg/Day): Total Basal
Description: as for outcome 14
Time Frame: At week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units/(kilogram) kg/day
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 144 | 144
Units/(kilogram) kg/day | 0.37 (0.19) | 0.39 (0.17)

18. Secondary Outcome: Insulin Dose (Units/kg/Day): Total Bolus
Description: as for outcome 15
Time Frame: At week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units/kg/day
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 144 | 144
Units/kg/day | 0.56 (0.23) | 0.57 (0.25)

19. Secondary Outcome: Insulin Dose (Units/kg/Day): Individual Meal Insulin Dose
Description: as for outcome 16
Time Frame: At week 16
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units/kg/day
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 144 | 144
Units/kg/day
  Breakfast | 0.17 (0.08) | 0.17 (0.09)
  Lunch | 0.19 (0.08) | 0.20 (0.09)
  Main evening meal | 0.20 (0.09) | 0.20 (0.09)

20. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: Number of treatment emergent adverse events were recorded from week 0 to week 16. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. TEAE was defined as an event that had an onset date on or after the first day of exposure to randomised treatment, and no later than seven days after the last day of exposure to randomised treatment.
Time Frame: From baseline (week 0) to 16 weeks after randomisation
Population: SAS which included all participants receiving at least one dose of randomised treatment.
Measure: Number; unit: Events
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Events | 285 | 263

21. Secondary Outcome: Number of Treatment Emergent Injection Site Reactions
Description: Number of treatment emergent injection site reactions were recorded from week 0 to week 16. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period.
Time Frame: From baseline (week 0) to 16 weeks after randomisation
Population: SAS which included all participants receiving at least one dose of randomised treatment.
Measure: Number; unit: Events
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Events | 0 | 0

22. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes Classified Both According to the American Diabetes Association (ADA) Definition and Novo Nordisk (NN) Definition: Overall
Description: ADA classification of hypoglycaemia as follows: 1) Severe: Requiring assistance to actively administer carbohydrate/glucagon/take other corrective actions. 2) Documented symptomatic: PG ≤3.9 mmol/L with symptoms. 3) Asymptomatic: PG ≤3.9 mmol/L without symptoms. 4) Probable symptomatic: No measurement with symptoms. 5) Pseudo-hypoglycaemia: PG >3.9 mmol/L with symptoms. 6) Unclassifiable. NN classification of hypoglycaemia as follows: 1) BG confirmed: PG <3.1 mmol/L with/without symptoms. 2) Severe or BG confirmed symptomatic: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with symptoms. 3) Severe or BG confirmed: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with/without symptoms. 4) Unclassifiable. Not able to self-treat-unclassifiable: Not able to self-treat but not classifiable as severe hypoglycaemia.
Time Frame: From baseline (week 0) to 16 weeks after randomisation
Population: SAS which included all participants receiving at least one dose of randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Episodes
  ADA: Severe | 1 | 0
  ADA: Documented symptomatic | 915 | 971
  ADA: Asymptomatic | 453 | 402
  ADA: Probable symptomatic | 0 | 0
  ADA: Pseudo-hypoglycaemia | 12 | 30
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 404 | 438
  NN: Severe or BG confirmed symptomatic | 316 | 347
  NN: Severe or BG confirmed | 404 | 438
  NN: Unclassifiable | 1 | 0

23. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes Classified Both According to the ADA Definition and NN Definition: Day Time Hypoglycaemic Episodes (00:01-05:59 - Both Inclusive)
Description: Number of treatment emergent day time hypoglycaemic episodes as per ADA and NN definitions were evaluated. ADA classification of hypoglycaemia as follows: 1) Severe: Requiring assistance to actively administer carbohydrate/glucagon/take other corrective actions. 2) Documented symptomatic: PG ≤3.9 mmol/L with symptoms. 3) Asymptomatic: PG ≤3.9 mmol/L without symptoms. 4) Probable symptomatic: No measurement with symptoms. 5) Pseudo-hypoglycaemia: PG >3.9 mmol/L with symptoms. 6) Unclassifiable. NN classification of hypoglycaemia as follows: 1) BG confirmed: PG <3.1 mmol/L with/without symptoms. 2) Severe or BG confirmed symptomatic: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with symptoms. 3) Severe or BG confirmed: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with/without symptoms. 4) Unclassifiable. Not able to self-treat-unclassifiable: Not able to self-treat but not classifiable as severe hypoglycaemia.
Time Frame: From baseline (week 0) to 16 weeks after randomisation
Population: SAS which included all participants receiving at least one dose of randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Episodes
  ADA: Severe | 0 | 0
  ADA: Documented symptomatic | 863 | 927
  ADA: Asymptomatic | 440 | 390
  ADA: Probable symptomatic | 0 | 0
  ADA: Pseudo-hypoglycaemia | 11 | 27
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 375 | 417
  NN: Severe or BG confirmed symptomatic | 292 | 327
  NN: Severe or BG confirmed | 375 | 417
  NN: Unclassifiable | 0 | 0

24. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes Classified Both According to the ADA Definition and NN Definition: Nocturnal Hypoglycaemic Episodes (00:01-05:59 - Both Inclusive)
Description: Number of treatment emergent nocturnal hypoglycaemic episodes as per ADA and NN definitions were evaluated. ADA classification of hypoglycaemia as follows: 1) Severe: Requiring assistance to actively administer carbohydrate/glucagon/take other corrective actions. 2) Documented symptomatic: PG ≤3.9 mmol/L with symptoms. 3) Asymptomatic: PG ≤3.9 mmol/L without symptoms. 4) Probable symptomatic: No measurement with symptoms. 5) Pseudo-hypoglycaemia: PG >3.9 mmol/L with symptoms. 6) Unclassifiable. NN classification of hypoglycaemia as follows: 1) BG confirmed: PG <3.1 mmol/L with/without symptoms. 2) Severe or BG confirmed symptomatic: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with symptoms. 3) Severe or BG confirmed: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with/without symptoms. 4) Unclassifiable. Not able to self-treat-unclassifiable: Not able to self-treat but not classifiable as severe hypoglycaemia.
Time Frame: From baseline (week 0) to 16 weeks after randomisation
Population: SAS which included all participants receiving at least one dose of randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Episodes
  ADA: Severe | 0 | 0
  ADA: Documented symptomatic | 49 | 43
  ADA: Asymptomatic | 10 | 10
  ADA: Probable symptomatic | 0 | 0
  ADA: Pseudo-hypoglycaemia | 1 | 3
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 28 | 19
  NN: Severe or BG confirmed symptomatic | 24 | 19
  NN: Severe or BG confirmed | 28 | 19
  NN: Unclassifiable | 0 | 0

25. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes Classified Both According to the ADA Definition and NN Definition: Hypoglycaemic Episodes From Start of Meal Until 30 Minutes
Description: Number of treatment emergent hypoglycaemic episodes as per ADA and NN definitions were evaluated during first 30-mins after start of meal. ADA classification of hypoglycaemia as follows: 1) Severe: Requiring assistance to actively administer carbohydrate/glucagon/take other corrective actions. 2) Documented symptomatic: PG ≤3.9 mmol/L with symptoms. 3) Asymptomatic: PG ≤3.9 mmol/L without symptoms. 4) Probable symptomatic: No measurement with symptoms. 5) Pseudo-hypoglycaemia: PG >3.9 mmol/L with symptoms. 6) Unclassifiable. NN classification of hypoglycaemia as follows: 1) BG confirmed: PG <3.1 mmol/L with/without symptoms. 2) Severe or BG confirmed symptomatic: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with symptoms. 3) Severe or BG confirmed: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with/without symptoms. 4) Unclassifiable. Not able to self-treat-unclassifiable: Not able to self-treat but not classifiable as severe hypoglycaemia.
Time Frame: From baseline (week 0) to 16 weeks after randomisation
Population: SAS which included all participants receiving at least one dose of randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Episodes
  ADA: Severe | 0 | 0
  ADA: Documented symptomatic | 6 | 8
  ADA: Asymptomatic | 1 | 1
  ADA: Probable symptomatic | 0 | 0
  ADA: Pseudo-hypoglycaemia | 0 | 0
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 2 | 3
  NN: Severe or BG confirmed symptomatic | 2 | 3
  NN: Severe or BG confirmed | 2 | 3
  NN: Unclassifiable | 0 | 0

26. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes Classified Both According to the ADA Definition and NN Definition: Hypoglycaemic Episodes From Start of Meal Until 1 Hour
Description: Number of treatment emergent hypoglycaemic episodes as per ADA and NN definitions were evaluated during first 1 hour after start of meal. ADA classification of hypoglycaemia as follows: 1) Severe: Requiring assistance to actively administer carbohydrate/glucagon/take other corrective actions. 2) Documented symptomatic: PG ≤3.9 mmol/L with symptoms. 3) Asymptomatic: PG ≤3.9 mmol/L without symptoms. 4) Probable symptomatic: No measurement with symptoms. 5) Pseudo-hypoglycaemia: PG >3.9 mmol/L with symptoms. 6) Unclassifiable. NN classification of hypoglycaemia as follows: 1) BG confirmed: PG <3.1 mmol/L with/without symptoms. 2) Severe or BG confirmed symptomatic: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with symptoms. 3) Severe or BG confirmed: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with/without symptoms. 4) Unclassifiable. Not able to self-treat-unclassifiable: Not able to self-treat but not classifiable as severe hypoglycaemia.
Time Frame: From baseline (week 0) to 16 weeks after randomisation
Population: SAS which included all participants receiving at least one dose of randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Episodes
  ADA: Severe | 0 | 0
  ADA: Documented symptomatic | 43 | 41
  ADA: Asymptomatic | 17 | 17
  ADA: Probable symptomatic | 0 | 0
  ADA: Pseudo-hypoglycaemia | 1 | 0
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 24 | 24
  NN: Severe or BG confirmed symptomatic | 20 | 20
  NN: Severe or BG confirmed | 24 | 24
  NN: Unclassifiable | 0 | 0

27. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes Classified Both According to the ADA Definition and NN Definition: Hypoglycaemic Episodes From Start of Meal Until 2 Hours
Description: Number of treatment emergent hypoglycaemic episodes as per ADA and NN definitions were evaluated during first 2 hours after start of meal. ADA classification of hypoglycaemia as follows: 1) Severe: Requiring assistance to actively administer carbohydrate/glucagon/take other corrective actions. 2) Documented symptomatic: PG ≤3.9 mmol/L with symptoms. 3) Asymptomatic: PG ≤3.9 mmol/L without symptoms. 4) Probable symptomatic: No measurement with symptoms. 5) Pseudo-hypoglycaemia: PG >3.9 mmol/L with symptoms. 6) Unclassifiable. NN classification of hypoglycaemia as follows: 1) BG confirmed: PG <3.1 mmol/L with/without symptoms. 2) Severe or BG confirmed symptomatic: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with symptoms. 3) Severe or BG confirmed: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with/without symptoms. 4) Unclassifiable. Not able to self-treat-unclassifiable: Not able to self-treat but not classifiable as severe hypoglycaemia.
Time Frame: From baseline (week 0) to 16 weeks after randomisation
Population: SAS which included all participants receiving at least one dose of randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Episodes
  ADA: Severe | 0 | 0
  ADA: Documented symptomatic | 126 | 147
  ADA: Asymptomatic | 33 | 39
  ADA: Probable symptomatic | 0 | 0
  ADA: Pseudo-hypoglycaemia | 3 | 4
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 66 | 81
  NN: Severe or BG confirmed symptomatic | 58 | 69
  NN: Severe or BG confirmed | 66 | 81
  NN: Unclassifiable | 0 | 0

28. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes Classified Both According to the ADA Definition and NN Definition: Hypoglycaemic Episodes From Start of Meal Until 4 Hours
Description: Number of treatment emergent hypoglycaemic episodes as per ADA and NN definitions were evaluated during first 4 hours after start of meal. ADA classification of hypoglycaemia as follows: 1) Severe: Requiring assistance to actively administer carbohydrate/glucagon/take other corrective actions. 2) Documented symptomatic: PG ≤3.9 mmol/L with symptoms. 3) Asymptomatic: PG ≤3.9 mmol/L without symptoms. 4) Probable symptomatic: No measurement with symptoms. 5) Pseudo-hypoglycaemia: PG >3.9 mmol/L with symptoms. 6) Unclassifiable. NN classification of hypoglycaemia as follows: 1) BG confirmed: PG <3.1 mmol/L with/without symptoms. 2) Severe or BG confirmed symptomatic: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with symptoms. 3) Severe or BG confirmed: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with/without symptoms. 4) Unclassifiable. Not able to self-treat-unclassifiable: Not able to self-treat but not classifiable as severe hypoglycaemia.
Time Frame: From baseline (week 0) to 16 weeks after randomisation
Population: SAS which included all participants receiving at least one dose of randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Episodes
  ADA: Severe | 0 | 0
  ADA: Documented symptomatic | 391 | 433
  ADA: Asymptomatic | 142 | 133
  ADA: Probable symptomatic | 0 | 0
  ADA: Pseudo-hypoglycaemia | 6 | 11
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 213 | 217
  NN: Severe or BG confirmed symptomatic | 176 | 181
  NN: Severe or BG confirmed | 213 | 217
  NN: Unclassifiable | 0 | 0

29. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes Classified Both According to the ADA Definition and NN Definition: Hypoglycaemic Episodes From 2 Hours (Exclusive) to 4 Hours (Inclusive) After Start of Meal
Description: Number of treatment emergent hypoglycaemic episodes as per ADA and NN definitions were evaluated from 2 hours to 4 hours after start of meal. ADA classification of hypoglycaemia as follows: 1) Severe: Requiring assistance to actively administer carbohydrate/glucagon/take other corrective actions. 2) Documented symptomatic: PG ≤3.9 mmol/L with symptoms. 3) Asymptomatic: PG ≤3.9 mmol/L without symptoms. 4) Probable symptomatic: No measurement with symptoms. 5) Pseudo-hypoglycaemia: PG >3.9 mmol/L with symptoms. 6) Unclassifiable. NN classification of hypoglycaemia as follows: 1) BG confirmed: PG <3.1 mmol/L with/without symptoms. 2) Severe or BG confirmed symptomatic: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with symptoms. 3) Severe or BG confirmed: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with/without symptoms. 4) Unclassifiable. Not able to self-treat-unclassifiable: Not able to self-treat but not classifiable as severe hypoglycaemia.
Time Frame: From baseline (week 0) to 16 weeks after randomisation
Population: SAS which included all participants receiving at least one dose of randomised treatment.
Measure: Number; unit: Episodes
Arm/Group | Faster aspart | NovoRapid
Number analyzed (Participants) | 150 | 150
Episodes
  ADA: Severe | 0 | 0
  ADA: Documented symptomatic | 265 | 286
  ADA: Asymptomatic | 109 | 94
  ADA: Probable symptomatic | 0 | 0
  ADA: Pseudo-hypoglycaemia | 3 | 7
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 147 | 136
  NN: Severe or BG confirmed symptomatic | 118 | 112
  NN: Severe or BG confirmed | 147 | 136
  NN: Unclassifiable | 0 | 0

ADVERSE EVENTS:
Time Frame: Run-in period up to 8 weeks, randomised treatment period up to 16 weeks
Description: All presented AEs are TEAEs, defined as an event that had an onset date on or after the first day of exposure to randomised treatment, and no later than seven days after the last day of exposure to randomised treatment. Results are based on the SAS which included all randomised participants exposed to at least one dose of randomised treatment.
Groups:
- NovoRapid: Run-in period: Participants received subcutaneous injections of NovoRapid thrice daily + insulin degludec once daily with or without metformin for 8 weeks. Insulin degludec dose was adjusted weekly by the investigator based on the mean of three pre-breakfast SMPG values measured on the last two days prior to and on the day of contact. If one of the SMPG values were below target (less than 4.0 mmol/L or 71 mg/dL) then the insulin degludec dose was adjusted according to the titration guideline specified in the protocol.
Arm/Group | NovoRapid: Run-in period | Faster aspart | NovoRapid
All-Cause Mortality (participants affected / at risk) | 0/331 | 0/150 | 0/150
Serious Adverse Events (participants affected / at risk) | 9/331 | 10/150 | 7/150
Other Adverse Events (participants affected / at risk) | 32/331 | 55/150 | 40/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NovoRapid: Run-in period (N=331) | Faster aspart (N=150) | NovoRapid (N=150)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric Polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Patella Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NovoRapid: Run-in period (N=331) | Faster aspart (N=150) | NovoRapid (N=150)
Diabetic retinopathy (Eye disorders) | 15 (16) | 22 (22) | 10 (10)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 14 (14)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 21 (21) | 15 (15)
Upper respiratory tract infection (Infections and infestations) | 22 (24) | 14 (15) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT04588259/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT04588259/SAP_001.pdf